CLINICAL TRIAL: NCT04998266
Title: Evaluation of Physical Capacities Within the Company and Effect of a Personalized Versus Traditional Training Program on the Quality of Life of Sedentary Employees: Randomized Controlled Trial
Brief Title: Evaluation of Physical Capacities Within the Company and Effect of a Personalized Versus Traditional Training Program on the Quality of Life of Sedentary Employees
Acronym: MOVING_LAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21CH116; 2021-A01511-40 (Other: ANSM)
Record Dates: First submitted 2021-08-03; First posted 2021-08-10 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Healthy Volunteers; Health
Keywords: sport; parallel; physiopathology; physical activity prescription; quality of life; exercise; Company
MeSH Terms: conditions — Motor Activity | interventions — World Health Organization

STUDY DESIGN:
Intervention Model Description: After first session evaluation, employees will be randomly assigned to one of the 2 followings groups: (1) group with traditional exercise (CLA) and group with adapted and personalized exercises (IND). The CLA group will perform exercises following World Health Organization (WHO) prescription while the IND group will perform strength, aerobic or flexibility exercises depending on their needs observed during the first assessment.
  Note that all session evaluations are investigated within the company of the participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized exercise group (IND) (Experimental): Group with adapted and personalized exercises (IND).The IND group will perform strength, aerobic or flexibility exercises depending on their needs observed during the first assessment.
  Interventions: Other: Performing on their needs
- Traditional exercise group (CLA) (Active Comparator): Group with traditional exercise (CLA). The CLA group will perform exercises following WHO (World Health Organization) prescription.
  Interventions: Other: Performing following WHO (World Health Organization)

INTERVENTIONS:
Other: Performing following WHO (World Health Organization) — The CLA group will perform exercises following WHO (World Health Organization) prescription
  Arms: Traditional exercise group (CLA)
Other: Performing on their needs — The IND group will perform strength, aerobic or flexibility exercises depending on their needs observed during the first assessment.
  Arms: Individualized exercise group (IND)

SUMMARY:
The practice of a physical activity, even moderate, plays an important role in the prevention and the management of the main chronic non-communicable diseases (cardiovascular diseases, certain cancers, diabetes, obesity, osteoporosis ...) as well as by improving psychological health. Several studies have shown that physical activity has a positive impact on the economy of companies via the reduction of absenteeism and the improvement of productivity. However, it seems important to individualize these recommendations in order to prescribe the best possible dose of physical activity for each individual. In this project, the investigators want to test the physical qualities of employees in order to prescribe the best possible dose of physical activity with the ultimate goal of improving quality of life.

The originality of this project is to evaluate physical capacities directly within the company of the participants instead of hospital unit.

DETAILED DESCRIPTION:
Physical activity (PA) is one of the major determinants of health. Indeed, the practice of a physical activity, even moderate, plays an important role in the prevention and the management of the main chronic non-communicable diseases (cardiovascular diseases, certain cancers, diabetes, obesity, osteoporosis ...) as well as by improving psychological health. The effects are beneficial regardless of age, gender and state of health. Moreover, in addition to the well-being of employees, several studies have shown that physical activity has a positive impact on the economy of companies via the reduction of absenteeism and the improvement of productivity. Today, the World Health Organization (WHO) prescribes 150 min of physical activity per week regardless of the person's profile (active employee, employee working in his office, construction worker, etc.).. In this project,the investigators therefore want to test the physical qualities of employees in order to prescribe the best possible dose of physical activity with the ultimate goal of improving quality of life.

ELIGIBILITY:
Inclusion Criteria

* Sedentary people
* Affiliate to health care organism
* Subject who gave their consent
* Employee of a company having accepted the terms of the study, as well as the agreement of the occupational physician

Exclusion Criteria:

* People with degenerative disease
* Cardiovascular trouble
* Subject who are not able to understand the proceeding of the study or to give their consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
SF-12 Score | At 6 months
  The primary outcome is a change in Short Form 12 (SF-12) score from baseline to 6 months of exercise intervention for the 2 groups (IND and CLA).
  Physical component scored between 0-72 Mental component scored between 0-70 For each component 0 mean a worse outcome

SECONDARY OUTCOMES:
Maximum oxygen consumption (VO2max in ml/kg/min) | At 6 months
  Maximum oxygen consumption (VO2max in ml/kg/min) during a sub-maximum exercise on an ergometric bike from baseline to 6 months of exercise intervention for both groups.
Power of the lower limbs of employees in watt (W) | At 6 months
  Measurement of the power (in W) developed during the realization of 2 sprints of a duration of 8 seconds interspersed by 2 minutes of recovery on the same ergonomic bicycle from baseline to 6 months of exercise intervention for both groups
Grip force in Newton (N) | At 6 months
  Grip force evaluated in Newton (N) by the dynamometer (or handgrip) from baseline to 6 months of exercise intervention for both groups.
Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-F) | At 6 months
  The perceived fatigue of employees will be assessed (from baseline to 6 months of exercise intervention for both groups) using the FACIT-F scale Scored between 0 and 52 A score below 34 means that the subject experiences significant fatigue in daily life, potentially impacting his quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: CLEMENT FOSCHIA, MD, Principal Investigator — CHU St-Etienne
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Mat Y, Casali C, Le Mat F, Feasson L, Foschia C, Gery M, Rossi J, Millet GY. Impact of a Self-Autonomous Evaluation Station and Personalized Training Algorithm on Quality of Life and Physical Capacities in Sedentary Adults: Randomized Controlled Trial. JMIR Form Res. 2024 Oct 4;8:e45461. doi: 10.2196/45461. PMID 39365990